CLINICAL TRIAL: NCT05004246
Title: Longitudinal Changes in Characteristics of COVID-19 Survivors and Their Long-term Follow-up Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Yichang Central People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Xiangya Hospital of Central South University (Other); Yunnan Provincial Infectious Disease Hospital (Other); WUHAN Number Seven HOSPITAL (Unknown); Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director of Department of Infectious Diseases, Tongji Hospital
Other Study IDs: TJ20210622
Record Dates: First submitted 2021-07-21; First posted 2021-08-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prognosis; Sequelae
Keywords: COVID-19; follow-up; consequences
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Follow-up study of Coronavirus disease 2019 (COVID-19) survivors has rarely been reported. We aimed to investigate longitudinal changes in the characteristics of COVID-19 survivors after discharge.

DETAILED DESCRIPTION:
From December 2019, coronavirus disease 2019 (COVID-19), caused by a β-coronavirus known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has spread across the globe. Numerous studies have been performed so far to investigate clinical characteristics, risk factors, potential treatment and pathogenesis of COVID-19. However, little information is available on the long-term prognosis and possible sequelae of COVID-19 survivors who have recovered and been discharged from hospital. Hence, the investigators conducted a prospective study to investigate the long-time prognosis and the possible sequelae of COVID-19 survivors. The investigators evaluated Demographic and clinical characteristics, laboratory and radiological findings,pulmonary function tests, electrocardiogram, complications as well as treatment and symptoms and signs of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with confirmed COVID-19 who have complete hospitalization data.

Exclusion Criteria:

Suspected cases of COVID-19.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll recovered patients with confirmed COVID-19 who were discharged from Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
symptoms and signs | 1-3years
  symptoms and signs will be collected.
SF-36 Questionnaire to the ability of Life | 1-3years
  Quality of Life will be assesed using the MOS item short from health survey（SF-36.Minimum value:0, Maximum value: 100. Higher scores mean a better outcome.
Mental quality | 1-3years
  Mental quality will be assessed using hospital anxiety and depression scale.Minimum value:0, Maximum value: 21. Higher scores mean a worse outcome.
laboratory findings,change from baseline for blood laboratory measures | 1-3years
  the change from baseline for laboratory examination （Hb in g/L, Leukocyte in /L, neutrophil count in /L，lymphocyte count in /L，Platelet count in /L，Creatinine in μmol/L, Bilirubin in mg/dL, ALP in U/L, γ-glutamyl transpeptidase in U/L，AST in U/L, ALT in U/L, Albumin in g/dL, triglycerides in mmol/L, total cholesterol in mmol/L，cardiac troponin I in ng/mL， myoglobin in ng/mL， brain natriuretic peptide precursors in pg/mL， lactate dehydrogenase in U/L, Creatine Kinase in U/L).
Radiological findings | 1-3years
  Radiological findings such as chest computed tomography will be assessed.
pulmonary function | 1-3years
  pulmonary function tests will be assessed.
Heart function | 1-3years
  electrocardiogram including arrhythmia,ST-T change and conduction block will be assessed.（they have no Units）
Abdominal ultrasound | 1-3years
  Abdominal ultrasound will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of infectious disease, Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided